CLINICAL TRIAL: NCT00688506
Title: Combined Sono-electro-magnetic Therapy for Treatment of Refractory Chronic Pelvic Pain Syndrome: A Prospective, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Combined Sono-electro-magnetic Therapy for Treatment of Refractory Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Thomas M. Kessler, MD, Department of Urology, University of Bern, 3010 Bern
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEK 292/07; 1492
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: Chronic pelvic pain syndrome; Neuromodulation; Brain effects; Neuroimaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Combined sono-electro-magnetic therapy
  Interventions: Device: combined sono-electro-magnetic therapy (Sonodyn Medico Star)
- 2 (Placebo Comparator): placebo therapy
  Interventions: Device: placebo therapy (Placebo Sonodyn Medico Star)

INTERVENTIONS:
Device: combined sono-electro-magnetic therapy (Sonodyn Medico Star) — twice a day for 10 minutes during 12 weeks
  Other Names: Sonodyn Medico Star
  Arms: 1
Device: placebo therapy (Placebo Sonodyn Medico Star) — twice a day for 10 minutes during 12 weeks
  Other Names: Placebo Sonodyn Medico Star device
  Arms: 2

SUMMARY:
Treatment of chronic pelvic pain syndrome (CPPS) is challenging for patients and physicians once conventional therapies fail.

We hypothesize that combined sono-electro-magnetic therapy can improve refractory CPPS in men. In addition, we postulate that combined sono-electro-magnetic therapy as well as placebo therapy has a significant effect on brain activity detectable by functional MRI.

ELIGIBILITY:
Inclusion Criteria:

* CPSS III
* symptomatic >3 months
* NIH-CPSI total score =/>15
* NIH-CPSI pain =/>8

Exclusion Criteria:

* post void residual >100mL
* urinary tract infection
* urethral stricture
* prostate cancer
* age <18 years
* claustrophobia
* pacemaker, neurostimulator, insulin / pain pump

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) | before treatment, after 6 and 12 weeks of treatment as well as 4 weeks after stop of treatment

SECONDARY OUTCOMES:
Brain activity assessed by functional MRI | before treatment, after 12 weeks of treatment
Comparison of MRI of CPPS patients versus MRI of age-/sex-matched controls of the local neuro-radiology MRI database | before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Kessler, MD, Principal Investigator — Department of Urology, University of Bern, 3010 Switzerland
Locations (1):
- Department of Urology, University of Bern, Bern, Switzerland

REFERENCES:
- [Derived] Kessler TM, Mordasini L, Weisstanner C, Juni P, da Costa BR, Wiest R, Thalmann GN. Sono-electro-magnetic therapy for treating chronic pelvic pain syndrome in men: a randomized, placebo-controlled, double-blind trial. PLoS One. 2014 Dec 29;9(12):e113368. doi: 10.1371/journal.pone.0113368. eCollection 2014. PMID 25546177